CLINICAL TRIAL: NCT04155112
Title: Hypocaloric Mediterranean Diet or Physical Activity to Lower Cardiometabolic Risk in Vulnerable Populations: the MeDiPA Study
Brief Title: Hypocaloric Mediterranean Diet or Physical Activity to Lower Cardiometabolic Risk
Acronym: MeDiPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: The National Association for Public Health, Norway (Other Government)
Responsible Party: Principal Investigator, Kari Anne Sveen, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/696
Record Dates: First submitted 2019-10-23; First posted 2019-11-07 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Overweight or Obesity; Obesity, Abdominal; Hypertension
Keywords: Hypertension; Lifestyle; Mediterranean diet; Physical activity; Weight loss
MeSH Terms: conditions — Overweight; Obesity; Obesity, Abdominal; Hypertension; Motor Activity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical activity (PA) (Experimental): For 6 months, the participants will be recommended to increase physical activity to ≥ 150 min of moderate intensity or ≥ 75 min of vigorous intensity aerobic PA (or an equivalent combination) and ≥ 2 days of resistance exercise a week. The participants will take part in supervised group classes, twice per week. Each participant will receive a heart rate monitor to bring home and to use while reporting activity via a physical activity diary.
  Interventions: Behavioral: Physical activity
- Hypocaloric Mediterranean diet (MeDi) (Experimental): For 6 months, the participants will be recommended to consume a diet for 5-10% body weight loss. This diet will be based on the Mediterranean diet pattern. For the 6 months of the intervention, the participants will weigh themselves weekly and report their progress to the investigator. Adaptations to the diet will be made to ensure the goal of 5-10% weight loss is achieved. Each participant will receive a scale to bring home and to use while reporting weight loss.
  Interventions: Behavioral: Hypocaloric Mediterranean diet
- Control (No Intervention): At baseline, participants will receive usual care, which consists of general information regarding the importance of lifestyle for BP. This information will not be reinforced throughout the study duration.

INTERVENTIONS:
Behavioral: Physical activity — Increased physical activity to the minimum recommended by health authorities (≥ 150 min of moderate intensity or ≥ 75 min of vigorous intensity aerobic PA (or an equivalent combination) and ≥ 2 days of resistance exercise a week).
  Other Names: PA
  Arms: Physical activity (PA)
Behavioral: Hypocaloric Mediterranean diet — Energy deficit to reach 5-10% weight loss within 6 months, based on the Mediterranean diet pattern.
  Other Names: MeDi
  Arms: Hypocaloric Mediterranean diet (MeDi)

SUMMARY:
The purpose of this randomized controlled trial is to test the effects of a hypocaloric Mediterranean diet or of physical activity in participants who take at least 2 antihypertensive drugs but do not reach blood pressure treatment goal.

This study is a randomized, controlled, single-center, parallel group trial with three arms: hypocaloric Mediterranean diet (MeDi), physical activity (PA), or control. The control group will receive usual care (no intervention). This study will not be blinded.

The interventions will last 6 months, while the study follow-up will last 12 months. Four study visits will take place: baseline, at 3 months, at 6 months, at 12 months. The primary outcome is change in mean 24-hour ambulatory systolic blood pressure and diastolic blood pressure among groups after 6 months of intervention. Secondary and exploratory outcomes include change in other measures of blood pressure, body composition, other markers of cardiometabolic disease, inflammation markers, safety outcomes, and quality of life, among others.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18 - 70 years
* Taking ≥ 2 antihypertensive drugs (includes combination therapy)
* Office SBP ≥ 140mmHg and/or DBP ≥ 90mmHg on two occasions
* BMI 25 - 40 kg/m2
* Waist circumference ≥ 88 cm (women) or ≥ 102 cm (men)
* Sedentary lifestyle (< 150 minutes/week of moderate intensity physical activity)
* Weight stable (± 5 kg in the last 6 months)
* Not on a weight loss diet
* Willing to comply to an intervention of either a hypocaloric Mediterranean diet or physical activity (or control) for 6 months

Exclusion Criteria:

* Unable to provide informed consent
* Pregnant or lactating
* Office BP ≥ 160/100 mmHg
* Diabetes mellitus type 1
* History of cardiovascular disease (including uncompensated heart failure, recent infarction or stroke in the last 6 months, severe arrhythmia, heart failure or unstable angina pectoris)
* Chronic kidney disease stages 4 or 5
* Cancer in the last 5 years
* Changes in concurrent medication (anti-hypertensives, anti-diabetics, lipid-lowering drugs) in the last 3 months
* Regular use of oral corticosteroids in excess of 5 mg prednisolone (or equivalent) during the last month
* Use of GLP-1 analogues for < 1 year
* Drug or alcohol abuse
* Eating disorders or severe dietary restrictions
* Impediments to physical activity at recommended levels due to musculoskeletal and other conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour ambulatory SBP among subjects, after 6 months. | Baseline to 6 months
  24-hour ambulatory blood pressure will be measured with a device that allows free-living.
  Change = (6 month measurement - baseline measurement).
Change in 24-hour ambulatory DBP among subjects, after 6 months. | baseline to 6 months
  24-hour ambulatory blood pressure will be measured with a device that allows free-living.
  Change = (6 month measurement - baseline measurement).

SECONDARY OUTCOMES:
Change in other measures of blood pressure, within and among subjects, after 6 and 12 months. | Baseline to 6 months, baseline to 12 months
  Blood pressure will be measured with 24-hour ambulatory blood pressure monitors and in-office. Other measures of blood pressure include daytime blood pressure, nighttime blood pressure, and office systolic and diastolic blood pressure.
  Change = (6 or 12 month measurement - baseline measurement)
Change in body composition, within and among subjects, after 6 months. | Baseline to 6 months
  Office measures of body composition will include weight, waist and hip circumferences, BMI, waist-to-hip ratio, and bioimpedance analysis (BIA). Additional measures of body composition will be acquired via Dual-energy X-ray absorptiometry (DXA), including fat mass, fat-free body mass, visceral adipose tissue, subcutaneous adipose tissue, and bone mineral content and density.
  Change = (6 month measurement - baseline measurement)
Change in markers of cardiometabolic risk, within and among subjects, after 6 and 12 months. | Baseline to 6 months, baseline to 12 months
  Cardiometabolic risk factors (including measures of glucose regulation, blood lipids, NORRISK 2 score, metabolic syndrome) will be measured via blood samples and additional clinical parameters.
  Change = (6 or 12 month measurement - baseline measurement)
Change in inflammation markers, within and among subjects, after 6 and 12 months. | Baseline to 6 months, baseline to 12 months
  Inflammation markers will be measured via blood tests (including CRP and differential leucocyte count).
  Change = (6 or 12 month measurement - baseline measurement)
Change in safety outcomes, within and among subjects, after 6 and 12 months. | Baseline to 6 months, baseline to 12 months
  Safety outcomes will be measured via blood tests (including hematology, kidney, liver, and thyroid markers).
  Change = (6 or 12 month measurement - baseline measurement)

OTHER OUTCOMES:
Change in quality of life, within and among subjects, after 3, 6 and 12 months. | Baseline to 6 months, baseline to 12 months
  Quality of life will be measured via the EQ-5D questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Anne Sveen, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Aker, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No